CLINICAL TRIAL: NCT03267602
Title: Role of Sleep Apnea in the Neuropsychological Function in Down Syndrome People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201208075RIC
Record Dates: First submitted 2017-08-17; First posted 2017-08-30 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Continuous Positive Airway Pressure (CPAP) Therapy (Experimental)
  Interventions: Device: CPAP

INTERVENTIONS:
Device: CPAP — If following patients are suffering from sleep apnea and agree to receive treatment,
  1. older than 18 years, AHI> 15 and present obvious symptoms or
  2. less than 18 years, AHI still> 5 after tonsillectomy and present obvious symptoms.
  Investigators will process CPAP treatment for 3 months, and do neuropsychological assessment and sleep examination after treatment for 6 months.

SUMMARY:
This is the first study about Neuropsychological function and OSAS in Taiwan. Although the correlation between OSAS and neuropsychological abnormalities had been reported, it is worth to understand more about the detailed domains that involved in our cohort. After this, investigators can dissect the cause of mental retardation in DS and help for further treatment strategies.

DETAILED DESCRIPTION:
Down Syndrome (DS) is the most common cause of mental retardation with incidence of 1 in 848 (Lin, Hu et al. 1991). Although prenatal Down syndrome and Amniocentesis had been applied for years, in the survey of 2005, current birth incidence of DS is 1.6 in 10,000 live birth, meaning a 30-50 new cases per year (Jou, Kuo et al. 2005). Patients with DS will have multisystemic manifestations including short stature, mental retardation, dysmorphism, congenital heart disease, congenital anomaly of gastrointestinal and genitourinary tract, abnormal endocrine function, leukemia and leukemoid reaction. Beside mental retardation, other anomalies could be treated or controlled by current medical care. The IQ of DS is around 20-80 with significant cognitive, language, and behavior problems (Dierssen, Ortiz-Abalia et al. 2006).

In addition, obstructive sleep apnea syndrome (OSAS) had been observed in DS people with prevalence about 45-79% in the literature (de Miguel-Diez, Villa-Asensi et al. 2003; Dyken, Lin-Dyken et al. 2003; Shott, Amin et al. 2006; Fitzgerald, Paul et al. 2007), which is much higher than the 1-3% prevalence rate in general population (Holmes 1993; Gislason and Benediktsdottir 1995). The reasons of DS people prone to have OSAS are due to the combination of anatomical and physiological factors. In DS people, facial dysmorphism (midfacial hypoplasia, mandibular hypoplasia), macroglossia, small hypopharynx, pharyngeal hypotonia, tonsil and adenoid enlargement, obesity, laryngomalacia, and tracheomalacia contributed to upper airway obstructions in DS people (Trois, Capone et al. 2009; Pandit and Fitzgerald 2012). In addition, DS people has increased incidence of lower respiratory tract diseases including gastroesophageal reflux, immunological dysfunction, tracheal bronchus, airway malacia, congenital heart disease, and pulmonary hypoplasia, which will predispose to OSAS. While growing up, DS people still have generalized hypotonia with increasing risk of developing hypothyroidism and obesity, which are also risk factors for OSAS (Trois, Capone et al. 2009).

It has been noted that sleep disordered breathing is associated with neurocognitive deficit, particularly of memory, learning, attention, hyperactivity, executive functioning, cognitive capacity, and poor school performance (Beebe 2006; Pandit and Fitzgerald 2012). And a number of studies have reported improved attention, executive functioning, analytical thinking, verbal functioning, memory and academic progress at 6-12 months post- adenotonsillectomy (Chervin, Ruzicka et al. 2006). In DS, study demonstrated that a higher number of apneic episodes on polysomnography was correlated to the decreased visuoperceptual skill in DS (Andreou, Galanopoulou et al. 2002). Similarly, presence of snoring in DS was associated with a much higher rate of disruptive school behavior than without snore (Carskadon, Pueschel et al. 1993). Although learning disability and memory defect had been globally known in DS, the behavior, cognitive, and developmental impairment caused by OSAS is especially concerning because it might adversely affect their ability, even the social adaptation (Rihtman, Tekuzener et al. 2010) . Therefore, investigators would like to know the correlation between severity of OSAS and Neurocognitive and behavior in DS people in Taiwan. Also, investigators would like to follow the Neurocognitive and behavior changes in those who had been treated for OSAS, including tonsillectomy or Bilevel Positive Airway Pressure.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with Down's syndrome by chromosome test, over 6 years old and IQ> 40.
2. Participants and caregiver who are willing and comply with study.

Exclusion Criteria:

1. Known to have uncontrolled heart, stomach, kidney or neurological / psychiatric disorders.
2. Cannot comply with study。

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Assessed the sleep apnea level with Apnoea-Hypopnoea Index (AHI) score. | 3 months
Assessed neuropsychological functions with Wechsler Preschool and Primary Scale of Intelligence (WPPSI-R) vocabulary subdomain score. | 3 months

SECONDARY OUTCOMES:
Assessed the memory domain that subtest of Sentence (WPPSI-R) . | 3 months
Assessed the memory domain that forward memory (Leiter International Performance Scale-Revised) . | 3 months
Evaluation of participants's Visuospatial functions with Geometric Design (WPPSI-R). | 3 months
Evaluation of participants's Visuospatial functions with Block Design (WPPSI-R). | 3 months
The Executive domain was assessed with TOWER (Developmental NEuroPSYchological Assessment, NEPSY) | 3 months
Assessed the Language domain with Vocabulary subtest | 3 months
Assessed the Sensorimotor domain with Visuomotor Precision-train and car | 3 months
Measurement the effectiveness of therapy before and after treatment with Apnoea-Hypopnoea Index (AHI). | 12 months
Measurement the effectiveness of therapy before and after treatment with Oxygen Desaturation Index (ODI). | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ni-Chung Lee, M.D, Ph.D, Principal Investigator — National Taiwan University Hospital